CLINICAL TRIAL: NCT04376606
Title: Changes of Left Atrial Function and Quality of Life After Transcatheter Closure of Left Atrial Appendage in Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruiqin xie (Other)
Responsible Party: Sponsor-Investigator, Ruiqin xie, director of cardiology department, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XieruiqindoctorLAAC
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; left atrial appendage closure; left atrial function; quality of life
MeSH Terms: conditions — Atrial Fibrillation | interventions — Left Atrial Appendage Closure; Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: A total of 105 patients with persistent atrial fibrillation(AF), who are persistented more than one year and planned to undergo surgical treatment, will be allocated into two groups. These patients will receive left atrial appendage closure, radiofrequency ablation under the guidance of 3D mapping and left atrial appendage closure combined with radiofrequency ablation, respectively (allocation ratio, 1:1:1)
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers will participate in the operation to record operative parameters such as LA pressure. Other researchers including follow-up personnel and the ultrasonic data analyst are uninformed about the random situation of the patients (patient information is recorded according to the random number. Random numbers corresponding to the random allocation list are stored in the research center. After follow-up of the last patient is completed, the random allocation list is published by the random number designer; and the designer does not participate in the data collection and statistics.)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Left atrial appendage closure group (Experimental)
  Interventions: Procedure: Left atrial appendage closure
- Radiofrequency ablation group (Experimental)
  Interventions: Procedure: Radiofrequency ablation
- LAAC combined with radiofrequency ablation group (Experimental)
  Interventions: Procedure: LAAC combined with radiofrequency ablation group

INTERVENTIONS:
Procedure: Left atrial appendage closure — Left atrial appendage closure is performed using a single endocardial plug devices guided by fluoroscopic guidance and transesophageal echocardiography
  Arms: Left atrial appendage closure group
Procedure: Radiofrequency ablation — Each patient with persistent AF receives circumferential pulmonary vein isolation under the 3D electro-anatomical mapping system , and no additional ablation is performed in the extrapulmonary sites unless the patient is diagnosed with atrial flutter before the operation.
  Arms: Radiofrequency ablation group
Procedure: LAAC combined with radiofrequency ablation group — Each patient received the same group of patients with simple radiofrequency ablation radiofrequency ablation treatment at the same time, the transcatheter occlusion of left atrial appendage opening
  Arms: LAAC combined with radiofrequency ablation group

SUMMARY:
A total of 105 (AF) patients with atrial fibrillation are scheduled to undergo surgery and will be divided into three groups. Left atrial appendage occlusion ((LAAC)), radiofrequency ablation guided by three-dimensional mapping and LAAC combined with radiofrequency ablation were performed respectively (allocation ratio 1:1:1). All patients were examined by real-time three-dimensional and two-dimensional ultrasound before operation and 3, 6 and 12 months after operation, and the (LA) function of left atrium was measured. All ultrasound data will be stored and the professional director of the ultrasound room will be invited to conduct quantitative analysis. Ultrasonic examination indexes include: anterior and posterior diameter of left atrium, left atrial ejection fraction and so on. All patients underwent transesophageal echocardiography before and 3 months after operation. The results were interpreted by 2 experienced ultrasound doctors to measure the presence of left atrial thrombus, residual shunt and device-related thrombus. Blood samples were taken to detect B-type natriuretic peptide before operation, 1 day, 3-6 months and 12 months after operation. All patients underwent 6-minute walking test and quality of life score before operation and 3, 6 and 12 months after operation. At the same time, the thickness of crest in all patients was measured during operation. This study will clarify the changes of left atrial function and quality of life in patients with atrial fibrillation after LAAC. In addition, this study also observed the effect of radiofrequency ablation combined with LAAC on left atrial function and evaluated whether one-stop surgery was superior to simple occlusion or ablation, and the above results were analyzed. The patients were followed up for an average of one year, and the changes of left atrial function, quality of life and embolic events were analyzed.

ELIGIBILITY:
Inclusion Criteria:

sustained AF attack occurred in patients with a duration of more than one year, patients taking class I and class III antiarrhythmic drugs could not prevent AF, patients younger than 80 years old， Cha2ds2-vasc score ≥2, not suitable for long-term oral anticoagulant drugs.

Exclusion Criteria:

Patients with a history of atrial thrombosis or valvular heart disease (moderate or severe valve stenosis or severe valve regurgitation), patients undergoing prosthetic heart valve replacement, pregnant women, patients with previous liver and kidney diseases, malignant tumors or blood system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Left atrial function of postoperative left atrial appendage occlusion detected | 1-12 months
  Transthoracic echocardiography
6-minute walking test | 1-12 months
  quality of life assessed
quality of life score test | 1-12 months
  quality of life assessed

SECONDARY OUTCOMES:
residual shunt and DRT after transcatheter closure of left atrial appendage detected | 1-12 months
  Transesophageal echocardiography
B natriuretic peptide assessed | 1-12 months
  Blood samples are extracted in all patients to detected

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China